CLINICAL TRIAL: NCT00356265
Title: Alpha-Adrenoceptor Vascular Function In Chronic Kidney Disease Focus On The Role Of Endothelial Nitric Oxide
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Futility: Impossible to recruit enough hypertensive participants to match Chronic Kidney Disease (CKD) participants on needed parameters.
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Crystal A. Gadegbeku, Associate Professor of Medicine, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUM 00000261; 5R33DK071222 (NIH)
Record Dates: First submitted 2006-07-24; First posted 2006-07-25 (Estimated); Results first posted 2018-01-23 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2017-12

CONDITIONS: Chronic Kidney Disease; Hypertension
Keywords: Blood Pressure Nitric Oxide; L-NMMA; Phenylephrine; Vasoreactivity; Blood Pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hypertension

STUDY DESIGN:
Intervention Model Description: All three groups will have the same intervention

ARMS (3):
- CKD (Experimental)
  Interventions: Drug: Procedure: Regional phenylephrine arterial infusion
- Hypertension group (Active Comparator)
  Interventions: Drug: Procedure: Regional phenylephrine arterial infusion
- Normotensive group (Active Comparator)
  Interventions: Drug: Procedure: Regional phenylephrine arterial infusion

INTERVENTIONS:
Drug: Procedure: Regional phenylephrine arterial infusion

SUMMARY:
The purpose of this study is to learn more about why most patients with early stages of kidney disease have high blood pressure.

We know the body produces natural substances that cause blood vessels to open wider to carry more blood when needed. An example is during exercise. Other natural substances cause blood vessels to get smaller and slow down blood flow when needed. An example is when people are cold. The balance between these substances is important. People with kidney disease and high blood pressure do not have the normal balance of these substances.

This study will include 3 groups of people, people with normal blood pressure, people with high blood pressure and people with kidney disease.

* Subjects will have a screening physical examination, including an ECG and laboratory tests
* Subjects with high blood pressure may not take their regular blood pressure medication for 3 weeks prior to the inpatient GCRC study
* Subjects will be given intra-arterial medications that will cause changes in the blood vessels during the in-patient study.

The study will then compare the responses of the three groups. A GFR test will be done to confirm the renal function of the group with chronic kidney disease.

These studies will provide insight into the mechanisms of the pathogenesis of enhanced α1 vasoreactivity in subjects with progressive renal disease. This will lay the groundwork for new strategies in the treatment and prevention of vascular disease among the rapidly growing group of individuals with CKD.

DETAILED DESCRIPTION:
Enhanced adrenergic vascular reactivity may significantly contribute to hypertension and the excessive cardiovascular disease burden in patients with chronic kidney disease (CKD). Nitric oxide (NO), a modulator of neurovascular function, may be linked to adrenergic vascular responsiveness. The central HYPOTHESIS is that the reduction in endothelial nitric oxide (NO) bioavailability contributes to the enhancement of α1-adrenoceptor vasomotor function in patients with CKD.

Specific Aims: In patients with mild to moderate CKD, compared to matched hypertensive and normotensive controls without CKD:

1. Determine if α1-adrenoceptor vasoreactivity is enhanced less by inhibition of endothelial NO
2. Determine whether α1-adrenoceptor vasoreactivity correlates with plasma levels of the endogenous NO inhibitor, asymmetrical dimethylarginine.

Methods: CKD will be confirmed by I125-iothalamate glomerular filtration rate. Regional α1-adrenoceptor vasoreactivity (sensitivity [EC50], reactivity [slope]) will be assessed by venous plethsymography using a graded intra-arterial infusion of the α1-adrenoceptor agonist, phenylephrine. Comparisons of vasoreactivity at baseline and during infusions of L-NMMA will be made between hypertensive non-diabetic subjects with glomerular filtrations rates between 30-70 ml/min age-, gender-, ethnicity- and % body fat-matched hypertensive and normotensive subjects with normal kidney function. In addition, plasma levels of the endogenous NO inhibitor, asymmetric dimethylarginine will be measured in the hypertensive subjects with and without CKD and compared to vasoreactivity.

Significance. These studies will provide insight into the mechanisms of the pathogenesis of enhanced α1 vasoreactivity in subjects with progressive renal disease.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women-18 to 55 years of age.
* There are three groups of volunteers.

  * Group A. People who are hypertensive with kidney disease. When not taking blood pressure medicines, blood pressure must have a systolic between 140-170 mmHg. Diastolic must be between 90-109 mmHg.Kidney function should be around half of normal. Urine protein must be no more than 1 gram in a 24-hour urine time period.
  * Group B. People who are hypertensive without kidney disease. Blood pressure must have a systolic between 140-170 mmHg. Diastolic must be between 90-109 mmHg. Kidney function should be normal. Normal amounts of protein in their urine.
  * Group C. People who are normotensive. Blood pressure must have a systolic below 131/mmHg. Diastolic must be below 81 mmHg. Kidney function should be normal. No more than normal amounts of protein in their urine.

Exclusion Criteria:

People with:

* Diabetes
* Lung disease
* Stomach disease
* Liver disease
* Blood vessel disease
* Heart disease
* Hereditary blood disorders
* Hematocrit (amount of red blood cells) less than 30%
* Current tobacco use
* Kidney disease who require dialysis
* Women who are pregnant or breastfeeding

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2006-07 (Actual); Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crystal A Gadegbeku, MD, Principal Investigator — Assistant Professor of Medicine, University of Michigan Health System, Department of Internal Medicine, Division of Nephrology
Locations (1):
- University of Michigan Hospital, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Three screen failures
Groups:
- Chronic Kidney Disease (CKD); Hypertension Group; Normotensive Group: Procedure: Regional phenylephrine arterial infusion
Period: Overall Study
Arm/Group | Chronic Kidney Disease (CKD) | Hypertension Group | Normotensive Group
Started | 7 | 2 | 6
Completed | 7 | 2 | 5
Not Completed | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Chronic Kidney Disease; Hypertension Group; Normotensive Group: Procedure: Regional phenylephrine arterial infusion
- Total: Total of all reporting groups
Arm/Group | Chronic Kidney Disease | Hypertension Group | Normotensive Group | Total
Number analyzed (Participants) | 7 | 2 | 6 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 7 | 2 | 6 | 15
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 4 | 7
  Male | 5 | 1 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 6 | 2 | 6 | 14
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 7 | 2 | 5 | 14
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 2 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: α1-adrenoceptor Vasoreactivity With L-NMMA
Description: Vasoreactivity is defined as Forearm blood flow, dose response curve; ml per minute per log of phenylephrine, or FABF ml/min/logPE;
  The x axis is the ml/min value and the y axis is the log Phenylephrine concentration.
Time Frame: up to 8 hours
Population: Based on the data from the 12 participants, and the early termination, no analysis was performed on the two hypertensive participants' data.
Measure: Mean (Standard Error); unit: ml/min x 1/log[PE]
Arm/Group | Chronic Kidney Disease | Normotensive Group
Number analyzed (Participants) | 7 | 5
ml/min x 1/log[PE]
  before L-NMMA infusion | -0.48 (0.10) | -0.22 (0.08)
  after L-NMMA infusion | -0.31 (0.09) | -0.16 (0.11)

2. Primary Outcome: α1-adrenoceptor Vasoreactivity With Endogenous ADMA
Time Frame: up to 8 hours
Population: The main goal of the study was to compare vasoreactivity across the three groups. Given the fact that we struggled to recruit matched hypertensive and normotensive control population, we were not able to achieve the goals of the study and therefore, ADMA levels were not measured.
Arm/Group | Chronic Kidney Disease | Hypertension Group | Normotensive Group
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were interviewed for safety follow up approximately 7 - 10 days after procedure.
Arm/Group | Chronic Kidney Disease | Hypertension Group | Normotensive Group
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/2 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/2 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No